CLINICAL TRIAL: NCT02764788
Title: Auriculotherapy Treatment in Fibromyalgia
Acronym: Fib-Auric
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015/27; 2015-A01842-47 (Other: ANSM)
Record Dates: First submitted 2016-05-04; First posted 2016-05-06 (Estimated); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: Fibromyalgia
Keywords: Auriculotherapy
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Specific auriculotherapy (Experimental): Auriculotherapy on specific points with needles
  Interventions: Other: Specific auriculotherapy
- Non-specific auriculotherapy (Sham Comparator): Auriculotherapy on non-specific auriculotherapy points with needles
  Interventions: Other: non-specific auriculotherapy
- Seed auriculotherapy (Placebo Comparator): Auriculotherapy on non-specific auriculotherapy points with seeds
  Interventions: Other: seed auriculotherapy

INTERVENTIONS:
Other: Specific auriculotherapy — Specific auriculotherapy with needles
  Arms: Specific auriculotherapy
Other: non-specific auriculotherapy — non-specific auriculotherapy with needles
  Arms: Non-specific auriculotherapy
Other: seed auriculotherapy — non-specific auriculotherapy with seeds
  Arms: Seed auriculotherapy

SUMMARY:
Fibromyalgia (FM) is the most common cause of diffuse pain in the bones and joints, and one of the most frequent causes of referral to the pain management unit. It affects mainly women; they are referred by a rheumatologist, an internal medicine physician or by their family physician.

FM produces various degrees of disability and pain, and has an important impact on quality of life. Sleep disorders, fatigue and cognitive dysfunctions are almost always part of the clinical presentation. The wide range of symptoms and signs, the unknown etiology, the lack of efficacy of pharmacological treatments make management of FM a very difficult task. In France the consensus includes limitation of pharmacological treatment, encouraging physical rehabilitation and referring the patients to a specialized pain clinic where multidisciplinary management will be undertaken. In our hospital the investigators favor non pharmacological therapies and propose to the FM patients to learn relaxation and self-hypnosis, physical rehabilitation and use of trans cutaneous electrical neurostimulation.

Auriculotherapy (AT) is a complementary therapy, based on the idea that the ear is a microsystem which reflects the entire body, represented on the auricle, the outer portion of the ear. Mapping of the auricle has been described, according to the fact that pathology of different organs can induce specific changes in the auricle, for example color change or sensitivity. Treating specific areas, which somehow would be "connected" to the affected organ could also improve the functioning of the body or relieve pain. AT uses placement of needles at points tailored to the patient's pathology. Whatever the mechanisms involved, the effectiveness of ATis currently supported by randomized controlled trials. It is validated by WHO since 1987, mapped in an international nomenclature initially proposed by Nogier.

The investigators regularly use AT in FM patients in our pain management unit to alleviate symptoms as pain, sleep disorders, anxiety. The investigators established a clinical trial in this population to assess impact of FM (assessed with Fibromyalgia Impact Questionnaire) following 3 months of AT management (Primary Outcome). Sleep disorder, fatigue, anxiety and depression, cognitive and physical dysfunction are also evaluated as secondary outcomes. The remnant effect of AT is also evaluated, 3 month after the end of the treatment by the same tests.

ELIGIBILITY:
Inclusion Criteria:

* fibromyalgia (criteria from ACR)

Exclusion Criteria:

* history or existing of inflammatory rheumatims, lupus, systemic diseases that may explain the pain syndrom
* history or existing of severe psychiatric desorder
* history or existing of hemophilia
* with anticoagulant treatment
* local counterindication to auriculotherapy
* valvular prosthesis
* auriculotherapy during the last 12 months
* new psychotherpeutic treatment which interfer with auriculotherapy
* pregnancy
* breath feeding
* RMI for the next 5 months

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-04-27 (Actual); Primary Completion 2022-03-09 (Actual); Study Completion 2022-03-09 (Actual)

PRIMARY OUTCOMES:
Effect of otherapy on the health of patients with fibromyalgia syndrome | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Mireille Michel-Cherqui, MD, Principal Investigator — Hopital Foch
Locations (1):
- Hopital Foch, Suresnes, France

IPD SHARING:
Plan to Share IPD: No